CLINICAL TRIAL: NCT00505271
Title: Phase I/II Evaluation of Safety and Efficacy of Pathotropic Nanoparticles Bearing a Dominant Negative Cyclin G1 Construct (Rexin-G) as Intervention for Recurrent or Metastatic Breast Cancer
Brief Title: Safety and Efficacy Study Using Rexin-G for Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Epeius Biotechnologies (Industry)
Responsible Party: Erlinda M. Gordon, M.D., Epeius Biotechnologies Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C07-104
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Rexin-G; Gene Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — retrovector encoding mutant anti-cyclin G1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Escalating doses of Rexin-G will be given two or three times a week for four weeks, with a 2 week rest period
  Interventions: Genetic: Rexin-G

INTERVENTIONS:
Genetic: Rexin-G — Three patients will receive Rexin-G at Dose Level I. If 1 of 3 patients at Dose Level I develops a grade 3 or 4 adverse event (CTCAE Version 3.0) which appears to be related or possibly related to Rexin-G, then 3 additional patients will be enrolled at the same dose level. If at least 2 of the first 3, or 3 of 6 patients at Dose Level I develop a grade 3 to 4 adverse event which appears to be related or possibly related to Rexin-G, accrual into the study will be held.
  At any dose level, up to six patients may be enrolled if there is evidence of biological activity in the first three patients. Dose escalation may stop if there is impressive evidence of biological activity. An amendment would be submitted to allow further expansion of dose level based on impressive biological activity.

SUMMARY:
The goal of the adaptive trial design is to confirm the over-all safety of Rexin-G and to determine the optimal dosing regimen for Rexin-G that would document the significant clinical benefits required to support a Phase II registration protocol for recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
The clinical trial incorporates a Phase II component that will evaluate the efficacy of Rexin-G using an adaptive trial design. Each treatment cycle will be six weeks: four weeks of treatment and two weeks of rest. Unlike a standard Phase I protocol, eligible patients may have repeat cycles after the safety data and objective tumor response/s are recorded. Continued Rexin-G treatment will enable the targeted nanomedicine to catch up with tumor growth, halt disease progression, and reduce tumor burden. The treatment strategy is to achieve tumor control as quickly as safely possible. The goal of the adaptive trial design is to confirm the over-all safety of Rexin-G and to determine the optimal dosing regimen for Rexin-G that would document the significant clinical benefits required to support a Phase II registration protocol for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed recurrent or metastatic breast cancer that is refractory to standard chemotherapy and that is measurable.
2. Adequate hepatic function: Total bilirubin < 2.0 mg/dL (upper limit included); AST/ALT < 2x institutional norm; alkaline phosphatase < 2.5x upper limit of institutional norm unless the patient has extensive bone metastases. Patients with elevated alkaline phosphatase due to extensive liver disease will be excluded from study; albumin > 3.0 mg/dL. There must be no substantial ascites. PT and PTT must be within normal limits.
3. Performance status must be < 1 (ECOG 0-1) with a life expectancy of at least 3 months.
4. Hemoglobin > 9 gms%
5. Absolute granulocyte count > 1000/uL, and platelet count > 100,000/uL.
6. Serum creatinine of less than 1.5 mg%.
7. There must be no plans for the patient to receive further cancer therapy from the date of enrollment until the completion of the 6-week follow-up visit.
8. Accessibility of peripheral or central IV line
9. Age > 18 years
10. Patients will be off chemotherapy for a minimum of 4 weeks prior to initiation of therapy and should have recovered to Grade 1 or less toxicity.
11. The ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior malignancy, except for non-melanoma skin cancer, stage 1 breast cancer, CIS of cervix from which the patient has been disease-free for 5 years.
2. Woman who are pregnant or nursing
3. Fertile patients unless they agree to use barrier contraception (condoms and spermicide jelly) during the vector infusion period and for six weeks after infusion. Male patients must agree to use barrier contraception.
4. Patients who are transfusion dependent (more than one transfusion per month)
5. Patients with medical, psychiatric, or social conditions that would compromise successful adherence to this protocol.
6. Patient who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2010-07 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Clinical toxicity (DLT and MTD) as defined by patient performance status, toxicity assessment score, hematologic and metabolic profiles. | 24 months

SECONDARY OUTCOMES:
To identify an objective tumor response to Rexin-G | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sant P Chawla, M.D., Principal Investigator — Epeius Clinical Research Unit/Sarcoma Oncology Center; Howard W Bruckner, M.D., Principal Investigator — Bruckner Oncology
Locations (3):
- United States (3):
  - Epeius Clinical Research Unit, San Marino, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Bruckner Oncology, New York, New York